CLINICAL TRIAL: NCT00505011
Title: Study of the Influence of the GST, CYP and TP53 Gene Polymorphisms in the Risk of Graves' Disease and Its Outcome.
Brief Title: Genetic Polymorphisms Associated With Cigarette Smoking and Risk of Graves' Disease
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Other Study IDs: 17072007
Record Dates: First submitted 2007-07-18; First posted 2007-07-20 (Estimated); Last update posted 2007-07-20 (Estimated); Status verified 2007-07

CONDITIONS: Graves' Disease
Keywords: susceptibility; genes; environment; ophthalmopathy; outcome
MeSH Terms: conditions — Graves Disease; Disease Susceptibility; Eye Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Cigarette smoking is a well-recognized risk factor of Graves' disease and, particularly, Graves' ophthalmopathy. Hence, germline polymorphisms of detoxification genes and genes belonging to the major DNA repair/apoptosis pathways might have an important role in disease susceptibility. In addition, as some of these genes are regulated by thyroid hormones, they could affect the outcome of these patients. Our objective was to assess the influence of the GST, CYP and TP53 gene polymorphisms in the risk of Graves' disease and its outcome.

DETAILED DESCRIPTION:
Although the role of many polymorphisms of genes related to toxins' metabolism has been extensively investigated regarding the susceptibility to thyroid cancer, their influence in thyroid autoimmune diseases risk is still largely unknown. Hence, this study was designed to assess the influence of GSTT1, GSTM1, GSTP1, CYP1A1 and 72TP53 polymorphic inheritance on the susceptibility to Graves' disease and to its response to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Graves' disease patients

Min Age: 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1998 (Actual)
Dates: Start 1998-02; Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura S Ward, MD, PhD, Principal Investigator — State University of Campinas- UNICAMP